CLINICAL TRIAL: NCT00628251
Title: A Phase II, Open-Label, Randomised, Comparative, International Multicentre Study to Assess the Safety and Efficacy of Different Doses of AZD2281 Given Orally Twice Daily Versus Intravenous Liposomal Doxorubicin Given Monthly in Patients With Advanced BRCA1- or BRCA2-Associated Ovarian Cancer Who Have Failed Previous Platinum-based Chemotherapy
Brief Title: Dose-finding Study Comparing Efficacy and Safety of a PARP Inhibitor Against Doxil in BRCA+ve Advanced Ovarian Cancer
Acronym: ICEBERG 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00012
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Neoplasms
Keywords: Advanced ovarian cancer; BRCA1 protein; BRCA2 protein; Poly(ADP ribose) polymerases
MeSH Terms: conditions — Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — olaparib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): AZD2281 Oral 200 mg BID
  Interventions: Drug: AZD2281
- 2 (Active Comparator): Liposomal Doxorubicin
  Interventions: Drug: Liposomal Doxorubicin
- 3 (Experimental): AZD2281 Oral 400 mg BID
  Interventions: Drug: AZD2281

INTERVENTIONS:
Drug: AZD2281 — 400mg Oral twice daily
  Other Names: Olaparib
  Arms: 3
Drug: Liposomal Doxorubicin — 50mg/m2 Monthly Intravenous
  Other Names: Doxil®
  Arms: 2
Drug: AZD2281 — 200mg oral twice daily
  Arms: 1

SUMMARY:
The purpose of the study is to compare the efficacy and safety of 2 doses of drug AZD2281 against liposomal doxorubicin to see which is effective and well tolerated in treating patients with measurable BRCA1- or BRCA2-positive advanced ovarian cancer and who have failed previous platinum therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced ovarian cancer with positive BRCA1 or BRCA2 status
* Progressive or recurrent disease after platinum-based chemotherapy
* Measurable disease by RECIST

Exclusion Criteria:

* Previous anthracycline treatment
* Brain metastases
* Less than 28 days since last treatment used to treat the disease
* Considered a poor medical risk due to a serious uncontrolled disorder

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-07-30 (Actual); Primary Completion 2009-09-15 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Stan Kaye, BSc, MB, FRCP, FRCR, SMedSCi, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (24):
- United States (6):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Boca Raton, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, East Melbourne
  - Research Site, Melbourne, Parkville
  - Research Site, Randwick
- Research Site, Leuven, Belgium
- Germany (2):
  - Research Site, Cologne
  - Research Site, München
- Israel (3):
  - Research Site, Haifa
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Research Site, Szczecin, Poland
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Hospitalet deLlobregat
- Research Site, Lund, Sweden
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Penson RT, Valencia RV, Cibula D, Colombo N, Leath CA 3rd, Bidzinski M, Kim JW, Nam JH, Madry R, Hernandez C, Mora PAR, Ryu SY, Milenkova T, Lowe ES, Barker L, Scambia G. Olaparib Versus Nonplatinum Chemotherapy in Patients With Platinum-Sensitive Relapsed Ovarian Cancer and a Germline BRCA1/2 Mutation (SOLO3): A Randomized Phase III Trial. J Clin Oncol. 2020 Apr 10;38(11):1164-1174. doi: 10.1200/JCO.19.02745. Epub 2020 Feb 19. PMID 32073956
- [Derived] Matulonis UA, Penson RT, Domchek SM, Kaufman B, Shapira-Frommer R, Audeh MW, Kaye S, Molife LR, Gelmon KA, Robertson JD, Mann H, Ho TW, Coleman RL. Olaparib monotherapy in patients with advanced relapsed ovarian cancer and a germline BRCA1/2 mutation: a multistudy analysis of response rates and safety. Ann Oncol. 2016 Jun;27(6):1013-1019. doi: 10.1093/annonc/mdw133. Epub 2016 Mar 8. PMID 26961146
- [Derived] Ang JE, Gourley C, Powell CB, High H, Shapira-Frommer R, Castonguay V, De Greve J, Atkinson T, Yap TA, Sandhu S, Banerjee S, Chen LM, Friedlander ML, Kaufman B, Oza AM, Matulonis U, Barber LJ, Kozarewa I, Fenwick K, Assiotis I, Campbell J, Chen L, de Bono JS, Gore ME, Lord CJ, Ashworth A, Kaye SB. Efficacy of chemotherapy in BRCA1/2 mutation carrier ovarian cancer in the setting of PARP inhibitor resistance: a multi-institutional study. Clin Cancer Res. 2013 Oct 1;19(19):5485-93. doi: 10.1158/1078-0432.CCR-13-1262. Epub 2013 Aug 6. PMID 23922302
- [Derived] Yap TA, Carden CP, Kaye SB. Beyond chemotherapy: targeted therapies in ovarian cancer. Nat Rev Cancer. 2009 Mar;9(3):167-81. doi: 10.1038/nrc2583. PMID 19238149
- See also: CSR_Synopsis_D0810C00012.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=193&filename=CSR_Synopsis_D0810C00012.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 30 July 2008 and last patient on 3 March 2009 at 25 centres in 9 countries
Pre-assignment Details: 97 of 125 screened women with advanced BRCA 1/2 ovarian cancer who had chemotherapy were randomized
Groups:
- Olaparib 200 mg bd: Olaparib (AZD2281) 200 mg oral capsules twice daily
- Olaparib 400 mg bd: Olaparib (AZD2281) 400 mg oral capsules twice daily
- Liposomal Doxorubicin: Liposomal doxorubicin 50 mg/m2 intravenously every 4 weeks
Period: Randomised Part
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Started | 32 (Patients randomised) | 32 (Patients randomised) | 33 (Patients randomised)
Completed | 32 (Patients who received olaparib treatment) | 32 (Patients who received olaparib treatment) | 32 (1 of 33 patients did not receive Liposomal Doxorubicin. Patient voluntarily discontinued)
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Ongoing Initial Study Treatment at DCO
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Started | 32 (Patients who received treatment) | 32 (Patients who received treatment) | 32 (Patients who received Liposomal doxorubicin 50 mg/m2)
Discontinued Initial Study Treatment | 22 | 20 | 25
Crossover to Olaparib | 0 | 0 | 14 (Crossover dosage was 400 mg bd Olaparib)
Ongoing Crossover at DCO | 0 | 0 | 5
Discontinued Crossover | 0 | 0 | 9
Completed | 10 (Ongoing initial study treatment at primary data cut-off) | 12 (Ongoing initial study treatment at primary data cut-off) | 7 (Patients ongoing initial study treatment (Liposomal doxorubicin))
Not Completed | 22 | 20 | 25
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Condition under investigation worsened | 19 | 15 | 13
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Other reason | 0 | 1 | 6
Not completed — Other | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin | Total
Number analyzed (Participants) | 32 | 32 | 33 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (8.53) | 53.8 (8.77) | 54.3 (9.32) | 55.5 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 33 | 97
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity (Jewish ethnicity)
  Participants
    African-Caribbean | 0 | 0 | 1 | 1
    Ashkenazi Jewish | 8 | 10 | 11 | 29
    Sephardic Jewish | 0 | 0 | 2 | 2
    Not applicable | 20 | 21 | 19 | 60
    Other | 4 | 1 | 0 | 5
BRCA status [Number; unit: Participants]
  Deleterious BRCA1 mutation | 26 | 28 | 27 | 81
  Deleterious BRCA2 mutation | 6 | 4 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time to progression from the date of randomisation until the date of radiological assessment of progression per RECIST criteria or death (by any cause in the absence of progression)
Time Frame: Tumour assessment was to be assessed at screening, every 8 weeks during the study and at the withdrawal visit, up to 56 weeks. (Data cut-off for primary analysis of PFS: 15 September 2009)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants | 19 | 20 | 20
Statistical Analysis 1: Comparison: Olaparib 200 mg bd vs Olaparib 400 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 200 or 400 mg bd (n=64) versus liposomal doxorubicin (n=33). A hazard ratio < 1 favours olaparib; Test type: Superiority or Other; p = 0.6604, Regression, Cox — If the observed p-value for the combined olaparib groups is <0.02 (1-sided) then the result will be regarded as statistically significant; Cox proportional hazards model with factors for treatment, BRCA (1 or 2) and platinum sensitivity (sensitive=1 or resistant/refractory=0); Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.51 to 1.56]
Statistical Analysis 2: Comparison: Olaparib 200 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 200 (n=32) versus liposomal doxorubicin (n=33). A hazard ratio < 1 favours olaparib; Test type: Superiority or Other; p = 0.7794, Regression, Cox — An observed p-value of <0.005 (1-sided) will be regarded as statistically significant for a given pairwise comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI [0.48 to 1.74]
Statistical Analysis 3: Comparison: Olaparib 400 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 400 (n=32) versus liposomal doxorubicin (n=33). A hazard ratio < 1 favours olaparib; Test type: Superiority or Other; p = 0.6604, Regression, Cox — An observed p-value of <0.005 (1-sided) will be regarded as statistically significant for a given pairwise comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.45 to 1.62]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined according to RECIST. Complete response (CR) or partial response - (PR)- 30% decrease Patients with a best RECIST response of CR or PR had to have a confirmed response at least 28 days later.
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants
  Complete response | 0 | 0 | 0
  Number of Partial responders | 8 | 10 | 6
Statistical Analysis 1: Comparison: Olaparib 200 mg bd vs Olaparib 400 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 200 or 400 (n=64) versus liposomal doxorubicin (n=33); Test type: Superiority or Other; p = 0.1291, Regression, Logistic — 2-sided p-value; Analysis was performed using logistic regression with factors for treatment, BRCA status and platinum sensitivity; Odds Ratio (OR) = 2.27, 95% CI 2-sided [0.79 to 7.32] — An odds ratio >1 favoured olaparib
Statistical Analysis 2: Comparison: Olaparib 200 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 200 (n=32) versus liposomal doxorubicin (n=33); Test type: Superiority or Other; p = 0.3131, Regression, Logistic — 2-sided p-value; Analysis was performed using logistic regression with factors for treatment, BRCA status and platinum sensitivity; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.55 to 7.01] — An odds ratio >1 favoured olaparib
Statistical Analysis 3: Comparison: Olaparib 400 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 400 (n=32) versus liposomal doxorubicin (n=33); Test type: Superiority or Other; p = 0.1079, Regression, Logistic; The analysis was performed using logistic regression with factors for treatment, BRCA status and platinum sensitivity; Odds Ratio (OR) = 2.69, 95% CI 2-sided [0.81 to 9.76] — An odds ratio >1 favoured olaparib

3. Secondary Outcome: Disease Control Rate
Description: The number of patients with confirmed CR (disappearance of all target lesions) or PR (30% decrease in the sum of the longest diameter of target lesions ) or SD ( small changes ) >4 months, divided by the number of randomised patients
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants | 21 | 21 | 19

4. Secondary Outcome: Overall Duration of Response
Description: The duration of response was defined as time (months) from initial assessment of PR/CR until earliest date of objective progression or death. (Values may be underestimated as some patients had not progressed at final analysis so true duration is likely to be greater than that in database.)
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Population: Duration of response is analysed for patients experiencing a response.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Olaparib 200 mg bd + Olaparib 400 mg bd,: Olaparib (AZD2281) 200 or 400 mg oral capsules twice daily
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Olaparib 200 mg bd + Olaparib 400 mg bd, | Liposomal Doxorubicin
Number analyzed (Participants) | 8 | 10 | 18 | 6
Months | 5.95 [3.71 to NA] — The upper limit for the 95% CI was not reached. | 6.80 [5.52 to 7.39] | 6.24 [5.52 to 7.39] | 5.49 [4.67 to 9.13]

5. Secondary Outcome: Best Percentage Change in Tumour Size
Description: The percentage change (reduction) from baseline in the sum of the lengths of the longest diameter (LD) of the RECIST target lesions were objectively documented, regardless of whether the patient was still taking study medication
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Measure: Median (Full Range); unit: Percent change
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Percent change | -15.90 [-75.30 to 31.48] | -24.60 [-100.00 to 51.10] | -14.3 [-87.5 to 32.4]

6. Secondary Outcome: Best Percentage Change From Baseline in CA-125 Levels
Description: Best percentage change in cancer antigen 125 (CA-125) levels
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Measure: Median (Full Range); unit: Percent change
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 30 | 31 | 33
Percent change | -37.42 [-98.77 to 327.76] | -71.19 [-96.88 to 70.56] | -55.8 [-99.5 to 192.1]

7. Secondary Outcome: Confirmed RECIST Response and/or CA-125 Response
Description: The percentage of patients reporting a RECIST confirmed response and/or a CA-125 response (in the absence of progression). A CA-125 response was defined as a confirmed greater or equal to 50% reduction in CA-125.
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Measure: Number; unit: Percentage of participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Percentage of participants | 37.5 | 59.4 | 39.4

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from randomisation to date of death from any cause. Patients who had not died at time of analysis were censored at last date they were known to be alive. Median OS was not calculable for olaparib groups due to an insufficient number of deaths so the percentage of participants who died are shown along with 95% confidence intervals
Time Frame: At the time of the cut-off for the final analysis of overall survival (30 April 2010)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants | 9 | 11 | 13
Statistical Analysis 1: Comparison: Olaparib 200 mg bd vs Olaparib 400 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 200 or 400 (n=64) versus liposomal doxorubicin (n=33); Test type: Superiority or Other; p = 0.5781, Regression, Cox — 2-sided p-value; Analysis was performed using a Cox proportional hazards model with factors for treatment, BRCA status and platinum sensitivity; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.41 to 1.70] — A hazard ratio of <1 favoured olaparib
Statistical Analysis 2: Comparison: Olaparib 200 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 200 (n=32) versus liposomal doxorubicin (n=33); Test type: Superiority or Other; p = 0.3417, Regression, Cox — 2-sided p-value; [statistical method as in outcome 8, analysis 1]; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.27 to 1.55] — A hazard ratio of <1 favoured olaparib
Statistical Analysis 3: Comparison: Olaparib 400 mg bd vs Liposomal Doxorubicin; Analysis of olaparib 400 (n=32) versus liposomal doxorubicin (n=33); Test type: Superiority or Other; p = 0.9877, Regression, Cox — 2-sided p-value; [statistical method as in outcome 8, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.44 to 2.27] — A hazard ratio of <1 favoured olaparib

9. Secondary Outcome: Best Quality of Life (QoL) Response for Trial Outcome Index (TOI)
Description: Best HRQoL response using the TOI endpoint. Improvement was defined as a change from baseline of greater than or equal to +7. The TOI score ranges from 0-100.
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Population: Evaluable for TOI at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants
  Improved | 7 | 5 | 3
  No change | 10 | 10 | 11
  Worsened | 3 | 7 | 6
  Non-evaluable | 5 | 7 | 7

10. Secondary Outcome: Best QoL Response for Total Functional Analysis of Cancer Therapy - Ovarian (FACT-O)
Description: Best HRQoL response using the total FACT-O endpoint. Improvement was defined as a change from baseline of greater than or equal to +9.
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Population: Evaluable for FACT-O at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants
  Improved | 3 | 6 | 1
  No Change | 14 | 11 | 11
  Worsened | 3 | 5 | 7
  Non-evaluable | 5 | 7 | 8

11. Secondary Outcome: Best QoL Response for FACT-O Symptom Index (FOSI)
Description: Best HRQoL response using the FOSI endpoint. Improvement was defined as a change from baseline of greater than or equal to +3.
Time Frame: At the time that 57 PFS events had occurred (Data cut-off for primary analysis of PFS: 15 September 2009)
Population: Evaluable for FOSI at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Participants
  Improved | 5 | 4 | 3
  No change | 14 | 9 | 10
  Worsened | 1 | 9 | 7
  Non-evaluable | 5 | 7 | 7

12. Primary Outcome: Progression Free Survival (PFS)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Number analyzed (Participants) | 32 | 32 | 33
Months | 6.5 [5.5 to 10.1] | 8.8 [5.4 to 9.2] | 7.1 [3.7 to 10.7]

ADVERSE EVENTS:
Description: AEs reported = all events up to OS data cut-off. After PFS data cut-off, AEs only collected for olaparib and cross-over groups. The safety profile of these 2 groups at OS was consistent with that at time of PFS. One patient was recorded as crossing over to olaparib but not receiving cross-over treatment.
Arm/Group | Olaparib 200 mg bd | Olaparib 400 mg bd | Liposomal Doxorubicin
Serious Adverse Events (participants affected / at risk) | 5/32 | 6/32 | 5/32
Other Adverse Events (participants affected / at risk) | 32/32 | 32/32 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib 200 mg bd (N=32) | Olaparib 400 mg bd (N=32) | Liposomal Doxorubicin (N=32)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib 200 mg bd (N=32) | Olaparib 400 mg bd (N=32) | Liposomal Doxorubicin (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 | 11 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 6
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2 | 1
Dry Eye (Eye disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 19 | 25 | 18
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 19
Vomiting (Gastrointestinal disorders) | 11 | 16 | 10
Abdominal Pain (Gastrointestinal disorders) | 12 | 8 | 12
Constipation (Gastrointestinal disorders) | 9 | 6 | 12
Diarrhoea (Gastrointestinal disorders) | 8 | 12 | 10
Dyspepsia (Gastrointestinal disorders) | 5 | 7 | 7
Abdominal Distension (Gastrointestinal disorders) | 3 | 3 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 4 | 3
Flatulence (Gastrointestinal disorders) | 2 | 4 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 2
Ascites (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 2
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 2
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 2 | 0
Fatigue (General disorders) | 12 | 21 | 14
Asthenia (General disorders) | 6 | 11 | 4
Mucosal Inflammation (General disorders) | 0 | 0 | 7
Pyrexia (General disorders) | 1 | 4 | 4
Chills (General disorders) | 0 | 1 | 3
Oedema Peripheral (General disorders) | 2 | 3 | 2
Pain (General disorders) | 0 | 1 | 2
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 5 | 11 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2 | 2
Influenza (Infections and infestations) | 3 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3
Bronchitis (Infections and infestations) | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Intertrigo Candida (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 0
Tinea Pedis (Infections and infestations) | 0 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 2 | 0
Viral Infection (Infections and infestations) | 2 | 2 | 1
Body Temperature Increased (Infections and infestations) | 1 | 3 | 0
Weight Decreased (Infections and infestations) | 2 | 2 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 5 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Headache (Nervous system disorders) | 8 | 9 | 8
Dizziness (Nervous system disorders) | 2 | 7 | 3
Dysgeusia (Nervous system disorders) | 5 | 5 | 0
Neuropathy Peripheral (Nervous system disorders) | 2 | 3 | 2
Memory Impairment (Nervous system disorders) | 2 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 4 | 2
Anxiety (Psychiatric disorders) | 2 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 20
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 7 | 1
Hot Flush (Vascular disorders) | 4 | 1 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
The AEs reported include all events up to the OS data cut-off. After the PFS data cut-off, AEs were only collected for the olaparib and cross-over groups. The safety profile of these 2 groups at OS was consistent with that at the time of PFS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication of the study results may be made until publication of the results of the multi-centre study or 2 years after study completion, whichever is the sooner